CLINICAL TRIAL: NCT03853850
Title: Strengthening Babies Through Mobile Health
Brief Title: Using Mobile Phone Text Messaging System to Improve Exclusive Breastfeeding Rate in a Resource-poor Caribbean Island
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Public Hospital Roatan, Honduras (Unknown); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-19171
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participating mothers will receive mobile phone text messages during their babies' first 6 months of life. Messages will educate mothers on breastfeeding and proper infant feeding.
  Interventions: Behavioral: Mobile phone text messages

INTERVENTIONS:
Behavioral: Mobile phone text messages — From their babies' day of birth until 6 months of age, participating mothers will receive supportive and educational text messages to promote breastfeeding. Messages will be on benefits of breastfeeding, newborn hunger cues, proper latch technique, healthy infant feeding practice, and maternal self care. Messages will be sent regularly, initially several messages every day during the babies' first few weeks of life, then few messages every week. A total of 158 (***) messages will be sent. Messages will be sent in English or in Spanish depending on participant language preference.

SUMMARY:
This study will evaluate whether sending educational and supportive mobile phone text messages to mothers of infants, from babies' day of birth until 6 months of age, increases the rate of exclusive breastfeeding in Roatan, Honduras.

DETAILED DESCRIPTION:
Encouraging and educational text messages and animations were created based on barriers to breastfeeding found during preceding focus groups and a baseline survey. Messages were written in English and translated into Spanish, with back-translation to ensure accuracy. Mothers who plan to or are already breastfeeding will be recruited and invited to participate in the study in the post-partum ward after delivery at Public Hospital Roatán. Written informed consent will be obtained. Three animated videos will be shown to mothers at enrollment providing information regarding breastfeeding technique, breastfeeding encouragement and general breastfeeding information. SMS messages will start at time of enrollment and continue through six months after enrollment. Messages will be delivered through Telerivet, an SMS interactive platform designed to send the educational and motivational messages to mothers' cell phones.

The intervention group will be polled when infants turn two months, four months, and six months regarding their infant feeding practices through Telerivet via SMS messaging. The primary outcome of this study is exclusive breastfeeding at 2 months of age, as compared to the exclusive breastfeeding rate obtained in our baseline cross sectional survey. Exclusive breastfeeding will be defined as giving only mother's breastmilk in the 24 hours preceding the interview. Mothers will also be asked if they are breastfeeding at all, age of infant when they last gave breast milk, the incidence of diarrheal illness in the past two weeks, and any other foods / liquids given to infant.

ELIGIBILITY:
Inclusion Criteria:

* Recently delivered full term infants (>37 weeks gestation, less than 72 hours old)
* 18 years of age or older, or emancipated minor, or if parent able to consent if <18 years of age
* Intent to breastfeed
* Own a phone that can receive SMS messages
* Able to send SMS reply messages

Exclusion Criteria:

* Mothers who report they can not read in Spanish nor English

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 582 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding rate at 2 months of age | 2 months after date of enrollment
  Proportion of infants exclusive breastfeeding at 2 months of age. Exclusive breastfeeding defined as only breastmilk in the 24 hours preceding data collection

SECONDARY OUTCOMES:
Exclusive breastfeeding rate at 4 months of age | 4 months after date of enrollment
  Proportion of infants exclusively breastfeeding at 4 months of age. Exclusive breastfeeding defined as only breastmilk in the 24 hours preceding data collection
Exclusive breastfeeding rate at 6 months of age | 6 months after date of enrollment
  Proportion of infants exclusively breastfeeding at 6 months of age. Exclusive breastfeeding defined as only breastmilk in the 24 hours preceding data collection
Breastfeeding rate at 4 months of age | 4 months after date of enrollment
  Proportion of infants with any amount of breastfeeding at 4 months of age
Breastfeeding rate at 6 months of age | 6 months after date of enrollment
  Proportion of infants with any amount of breastfeeding at 6 months of age
Diarrheal disease at 2 months of age | 2 months after date of enrollment
  Diarrheal disease incidence at 2 months of age. Diarrheal disease defined as watery stool during 2 weeks preceding data collection
Diarrheal disease at 4 months of age | 4 months after date of enrollment
  Diarrheal disease incidence at 4 months of age. Diarrheal disease defined as watery stool during 2 weeks preceding data collection
Diarrheal disease at 6 months of age | 6 months after date of enrollment
  Diarrheal disease incidence at 6 months of age. Diarrheal disease defined as watery stool during 2 weeks preceding data collection
Infant feeding practice at 2 months of age | 2 months after date of enrollment
  Other types of food given during 24 hours preceding data collection at 2 months of age
Infant feeding practice at 4 months of age | 4 months after date of enrollment
  Other types of food given during 24 hours preceding data collection at 4 months of age
Infant feeding practice at 6 months of age | 6 months after date of enrollment
  Other types of food given during 24 hours preceding data collection at 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chantry, MD, Principal Investigator — University of California, Davis; Lisa Rasmussen, MD, Principal Investigator — University of California, Davis
Locations (1):
- Public Hospital Roatan, Coxen Hole, Roatan, Honduras

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03853850/Prot_SAP_000.pdf